CLINICAL TRIAL: NCT00449865
Title: A Multicenter, Double-Blind, Parallel Group, Placebo Controlled Study of Creatine in Subjects With Treated Parkinson's Disease (PD) Long Term Study (LS-1)
Brief Title: NET-PD LS-1 Creatine in Parkinson's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Karl Kieburtz, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS43128 NET-PD; CRC; U01NS043128 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; creatine; NET-PD; neuroprotection; PD
MeSH Terms: conditions — Parkinson Disease | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- creatine (Active Comparator)
  Interventions: Drug: creatine

INTERVENTIONS:
Drug: creatine — Creatine, a widely used dietary supplement is thought to improve exercise performance. In animal models and human studies, creatine has been shown to be well tolerated and may have some ability to protect brain cells.
  The study is comparing creatine 5 grams twice daily with placebo.
  Arms: creatine
Other: placebo — an inactive substance
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine if the nutritional supplement creatine slows the progression of Parkinson's disease over time.

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects nearly a million Americans, a number that will increase over the coming decades as the population ages. Symptoms of PD may include tremor, rigidity or stiffness of the limbs and trunk, slowness of movement, and impaired balance and coordination. These problems occur because as PD worsens, some of the brain cells that control body movement die.

This study will determine if creatine--an investigational compound--is able to slow the progression of PD. Creatine, a widely used dietary supplement is thought to improve exercise performance. In animal models and human studies, creatine has been shown to be well tolerated and may have some ability to protect brain cells.

In the NET-PD LS-1 study, 1,720 participants will be randomly assigned to receive either creatine or a placebo (inactive substance). Participation in this study lasts a minimum of 5 years and includes at least 9 follow-up clinic visits and at least 3 telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent and willing to commit to long-term follow-up
* PD (asymmetric features including slowness (bradykinesia) plus resting tremor and/or rigidity) within 5 years of diagnosis
* Treated/responsive to dopaminergic therapy (dopamine agonists or levodopa) for at least 90 days, but not more than 2 years.

Exclusion Criteria:

* Use of creatine 14 days prior to baseline or during the study
* History of known hypersensitivity or intolerability to creatine
* Any unstable or clinically significant condition that would impair the subject's ability to comply with long term study follow-up
* Other know or suspected causes of parkinsonism (e.g. metabolic, drug induced, etc.), or any significant features suggestive of a diagnosis of atypical parkinsonism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1741 (Actual)
Dates: Start 2007-03; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Kieburtz, MD, Principal Investigator — Coordination Center; Barbara Tilley, PhD, Principal Investigator — Statistics Center
Locations (50):
- United States (48):
  - University Of Alabama, Birmingham, 350 Sparks Center, 1720 7th Avenue South, Birmingham, Alabama
  - Barrow Neurological Clinics At, St Joseph's Hospital & Medical Center, 500 West Thomas Road Suite 720,, Phoenix, Arizona
  - Parkinson's & Movement Disorder Institute, 9940 Talbert Avenue, Suite 204,, Fountain Valley, California
  - University Of Southern California, Healthcare Consultation Building II, 1520 San Pablo Street Suite 3000, Los Angeles, California
  - University Of California San Francisco, Parkinson's Disease Clinic And Research Cen, 505 Parnassus Avenue M-798, San Francisco, California
  - The Parkinson's Institute, 675 Almanor Avenue, Sunnyvale, California
  - University Of Colorado Health Sciences Ctr, 4200 East 9th Avenue Campus Box C238, Department Of Clinical Pharmacy, Denver, Colorado
  - Neurodegenerative Disorders, 60 Temple Street Suite 8b, New Haven, Connecticut
  - VA Medical Center, 1601 Southwest Archer Road, Neurology Service (151), Gainesville, Florida
  - University Of Florida, Mcknight Brain Institute, 100 South Newell Drive Room L3-100, Gainesville, Florida
  - University Of Florida Jacksonville, 580 West 8th Street, Tower 1 8th Floor,, Jacksonville, Florida
  - University Of Miami, 1501 North West 9th Avenue Second Floor, Department Of Neurology D4-5, Miami, Florida
  - University Of South Florida, Movement Disorders Center, 5 Tampa General Circle Suite 410, Tampa, Florida
  - Emory University, Wesley Woods Health Center, 1841 Clifton Road NE Room 328, Atlanta, Georgia
  - Medical College Of Georgia, Movement Disorders Clinic, 1429 Harper Street HF 1121, Augusta, Georgia
  - Pacific Health Research Institute, 405 North Kuakini Street, Suite 1011,, Honolulu, Hawaii
  - Northwestern University, 710 North Lake Shore Drive, Chicago, Illinois
  - Rush University Medical Center, Department Of Neurological Sciences, 1725 West Harrison Suite 755,, Chicago, Illinois
  - Evanston Northwestern Healthcare, Department Of Neurology, 2100 Pfingsten Road Suite B110, Glenview, Illinois
  - Southern Illinois University School Of Medicine, PO Box 19645, Springfield, Illinois
  - Indiana University School Of Medicine, Outpatient Clinical Research Facility, 535 Barnhill Drive Room #150, Indianapolis, Indiana
  - University Of Kansas Medical Center, 3599 Rainbow Blvd, Department Of Neurology Mail Stop # 2012, Kansas City, Kansas
  - University Of Kentucky Clinical Research, C201 Kentucky Clinic, 740 South Limestone Street, Lexington, Kentucky
  - Ochsner Clinic Foundation, 1514 Jefferson Highway, Dept. Of Neurology 7th Floor, New Orleans, Louisiana
  - LSU Health Science Center Shreveport, 1501 Kings Highway, Room 3-436, Shreveport, Louisiana
  - University Of Maryland School Of Medicine, Department Of Neurology, 22 South Greene Street N4W46, Baltimore, Maryland
  - Johns Hopkins University, 601 North Caroline Street, Suite 5064, Baltimore, Maryland
  - Brigham & Women's Hospital, Neurology Department ASB2, 75 Francis Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, 330 Brookline Avenue Shapiro 809D, Boston, Massachusetts
  - University Of Michigan, 1500 E Medical Center Drive, B1 H202 Nuclear Medicine,, Ann Arbor, Michigan
  - Michigan State University, Department Of Neurology A217 Clinical Center, 138 Service Road, East Lansing, Michigan
  - Struthers Parkinson's Center, 6701 Country Club Drive,, Golden Valley, Minnesota
  - Washington University School Of Medicine, 660 South Euclid Avenue, Campus 8111,, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, One Medical Center Drive, 2 Buck Road, Lebanon, New Hampshire
  - UMDNJ Robert Wood Johnson Medical School, Dept Of Neurology Suite 6100, 125 Paterson Street, New Brunswick, New Jersey
  - SUNY Downstate Medical Center, 450 Clarkson Avenue, Department Of Neurology Box 1213, Brooklyn, New York
  - Northshore-LIJ Health System, The Feinstein Institute FPR Medical Research, 350 Community Drive Room,, Manhasset, New York
  - Duke University Medical Center, Duke Health Center At Morreene Road, 932 Morreene Road Room 213,, Durham, North Carolina
  - OHSU Oregon Health &Science University, Department Of Neurology, 3181 South West Sam Jackson Park Road, Portland, Oregon
  - Thomas Jefferson University, 1015 Chestnut Street Suite 520, Philadelphia, Pennsylvania
  - University of Pennsylvania; Pennsylvania Hospital, Penn Neurological Institute, 330 South Ninth Street, Philadelphia, Pennsylvania
  - Thomas Jefferson University/Lankenau Hospital, Lankenau Medical Building Suite 161 East, 100 Lancaster Avenue, Wynnewood, Pennsylvania
  - Medical University Of South Carolina, Charleston Memorial Hospital, 326 Calhoun Street Suite 308, Charleston, South Carolina
  - Vanderbilt University Medical Center, 2311 Pierce Avenue, Room 2217,, Nashville, Tennessee
  - University Of Texas Southwestern Med Ctr. At Dallas, 5323 Harry Hines Boulevard H1-108, Dallas, Texas
  - Baylor College Of Medicine, 6550 Fannin Suite 1801, Houston, Texas
  - University Of Vermont, Department Of Neurology , Given Building C-219, 89 Beaumont Avenue, Burlington, Vermont
  - University Of Virginia Neurology Fontaine, Department Of Neurology, 500 Ray C Hunt Drive, Charlottesville, Virginia
- Canada (2):
  - University Of Calgary Movement Disorders Program, Dept Of Clin Neurosciences Area 3 Neurology, 3350 Hospital DR NW Health Sciences Centre, Calgary, Alberta
  - University Of Alberta, 10230-111 Avenue Room 0601, Movement Disorders Clinic Glenrose Rehab Hospital, Edmonton, Alberta

REFERENCES:
- [Derived] Leehey M, Luo S, Sharma S, Wills AA, Bainbridge JL, Wong PS, Simon DK, Schneider J, Zhang Y, Perez A, Dhall R, Christine CW, Singer C, Cambi F, Boyd JT. Association of metabolic syndrome and change in Unified Parkinson's Disease Rating Scale scores. Neurology. 2017 Oct 24;89(17):1789-1794. doi: 10.1212/WNL.0000000000004572. Epub 2017 Sep 29. PMID 28972194
- [Derived] Wills AM, Li R, Perez A, Ren X, Boyd J; NINDS NET-PD Investigators. Predictors of weight loss in early treated Parkinson's disease from the NET-PD LS-1 cohort. J Neurol. 2017 Aug;264(8):1746-1753. doi: 10.1007/s00415-017-8562-4. Epub 2017 Jul 15. PMID 28712000
- [Derived] Augustine EF, Dorsey ER, Hauser RA, Elm JJ, Tilley BC, Kieburtz KK. Communicating with participants during the conduct of multi-center clinical trials. Clin Trials. 2016 Dec;13(6):592-596. doi: 10.1177/1740774516665596. Epub 2016 Aug 29. PMID 27573636
- [Derived] Wills AM, Perez A, Wang J, Su X, Morgan J, Rajan SS, Leehey MA, Pontone GM, Chou KL, Umeh C, Mari Z, Boyd J; NINDS Exploratory Trials in Parkinson Disease (NET-PD) Investigators. Association Between Change in Body Mass Index, Unified Parkinson's Disease Rating Scale Scores, and Survival Among Persons With Parkinson Disease: Secondary Analysis of Longitudinal Data From NINDS Exploratory Trials in Parkinson Disease Long-term Study 1. JAMA Neurol. 2016 Mar;73(3):321-8. doi: 10.1001/jamaneurol.2015.4265. PMID 26751506
- [Derived] Writing Group for the NINDS Exploratory Trials in Parkinson Disease (NET-PD) Investigators; Kieburtz K, Tilley BC, Elm JJ, Babcock D, Hauser R, Ross GW, Augustine AH, Augustine EU, Aminoff MJ, Bodis-Wollner IG, Boyd J, Cambi F, Chou K, Christine CW, Cines M, Dahodwala N, Derwent L, Dewey RB Jr, Hawthorne K, Houghton DJ, Kamp C, Leehey M, Lew MF, Liang GS, Luo ST, Mari Z, Morgan JC, Parashos S, Perez A, Petrovitch H, Rajan S, Reichwein S, Roth JT, Schneider JS, Shannon KM, Simon DK, Simuni T, Singer C, Sudarsky L, Tanner CM, Umeh CC, Williams K, Wills AM. Effect of creatine monohydrate on clinical progression in patients with Parkinson disease: a randomized clinical trial. JAMA. 2015 Feb 10;313(6):584-93. doi: 10.1001/jama.2015.120. PMID 25668262
- See also: NET PD website — http://www.parkinsontrial.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine: creatine monohydrate (10 gram /day)
Period: Overall Study
Arm/Group | Placebo | Creatine
Started | 867 | 874
Completed Year 1 | 802 (867 Expected at Year 1) | 822 (874 Expected at Year 1)
Completed Year 2 | 768 (867 Expected at Year 2) | 766 (874 Expected at Year 2)
Completed Year 3 | 719 (867 Expected at Year 3) | 715 (874 Expected at Year 3)
Completed Year 4 | 521 (679 Expected at Year 4) | 523 (686 Expected at Year 4)
Completed | 345 (478 Expected at Year 5) | 340 (477 Expected at Year 5)
Not Completed | 522 | 534
Not completed — Withdrawal by Subject | 110 | 110
Not completed — Lost to Follow-up | 36 | 37
Not completed — Physician Decision | 13 | 12
Not completed — Death | 31 | 40
Not completed — Protocol Violation | 8 | 7
Not completed — Study was stopped | 324 | 328

BASELINE CHARACTERISTICS:
Groups:
- Creatine: creatine 5 grams twice daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Creatine | Total
Number analyzed (Participants) | 867 | 874 | 1741
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.6) | 62.1 (9.7) | 61.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 305 | 618
  Male | 554 | 569 | 1123
Time since diagnosis, y [Mean (Standard Deviation); unit: years] | 1.6 (1.1) | 1.5 (1.1) | 1.5 (1.1)
Total Unified Parkinson's Disease Rating Scale (UPDRS) [Mean (Standard Deviation); unit: units on a scale] — The total UPDRS is the sum of parts I, II, and III. The possible range of the total UPDRS is from 0-176. Higher values indicate worse outcomes.
  units on a scale | 25.9 (11) | 26.5 (11.7) | 26.2 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: The Global Outcome Combined Information on Change From Baseline in Schwab England Activities of Daily Living, 39-Item Parkinson's Disease Questionnaire, Ambulatory Capacity, Symbol Digit Modalities, and Modified Rankin at 5 Years.
Description: All outcomes were coded such that higher scores indicated worse outcomes. Patients were ranked on each outcome and their ranks were summed (summed-ranks). Higher summed ranks (range, 5-4775) indicate worse outcomes. The mean summed ranks were compared by treatment group by a global statistical test (GST).
Time Frame: Change from baseline to 5 YEARS
Population: Intent-to-Treat sample: n = 955, participants randomized at least 5 years before July 2013 (time of planned interim analysis).
Measure: Mean (95% Confidence Interval); unit: summed-ranks
Groups:
- Creatine: creatine monohydrate (10 grams/day)
Arm/Group | Placebo | Creatine
Number analyzed (Participants) | 478 | 477
summed-ranks | 2360 [2249 to 2470] | 2414 [2304 to 2524]
Statistical Analysis 1: Comparison: Placebo vs Creatine; Test type: Superiority or Other; p = 0.45, Global Statistical Test; The global statistical test yielded t = -0.75 (2-sided p-value = .45, df=1865.8)

ADVERSE EVENTS:
Arm/Group | Placebo | Creatine
Serious Adverse Events (participants affected / at risk) | 347/867 | 315/874
Other Adverse Events (participants affected / at risk) | 687/867 | 698/874
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=867) | Creatine (N=874)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 9
Bradycardia (Cardiac disorders) | 4 | 0
Brugada syndrome (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 7
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 4
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 8 | 12
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 1 | 0
Factor V deficiency (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 5 | 2
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 15 | 14
Cyst (General disorders) | 0 | 2
Death (General disorders) | 2 | 5
Drug interaction (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 2
Pain (General disorders) | 9 | 4
Ulcer (General disorders) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 3
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 4 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 4 | 4
Clostridial infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Coccidioidomycosis (Infections and infestations) | 1 | 0
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 2 | 0
Groin abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Hip infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 1 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Oesophageal infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peridiverticulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 18 | 16
Pyelonephritis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 9 | 5
Urosepsis (Infections and infestations) | 4 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 11 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 12 | 10
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 4 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 4 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1
Catheterisation cardiac (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Investigation (Investigations) | 0 | 1
Medical observation (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 11
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 15
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 11 | 4
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 6
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial hypotension (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 3
Migraine (Nervous system disorders) | 1 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 4 | 4
Presyncope (Nervous system disorders) | 3 | 2
Sciatica (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Spinal cord disorder (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 15 | 12
Transient ischaemic attack (Nervous system disorders) | 6 | 4
Tremor (Nervous system disorders) | 2 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 3 | 2
Delusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Food aversion (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 3 | 3
Hallucination, visual (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Bladder disorder (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 2 | 3
Contracted bladder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 6 | 2
Renal colic (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 4 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Cystocele (Reproductive system and breast disorders) | 2 | 2
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Joint dislocation (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 4 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Angioplasty (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 3 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1
Benign tumour excision (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 2
Cholecystectomy (Surgical and medical procedures) | 0 | 3
Colporrhaphy (Surgical and medical procedures) | 0 | 1
Deep brain stimulation (Surgical and medical procedures) | 27 | 24
Heart valve replacement (Surgical and medical procedures) | 1 | 0
Hernia hiatus repair (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 5 | 2
Hysterectomy (Surgical and medical procedures) | 2 | 3
Joint arthroplasty (Surgical and medical procedures) | 1 | 5
Knee arthroplasty (Surgical and medical procedures) | 5 | 3
Large intestine anastomosis (Surgical and medical procedures) | 0 | 1
Meniscus operation (Surgical and medical procedures) | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 1
Prophylaxis of nausea and vomiting (Surgical and medical procedures) | 0 | 1
Prostatectomy (Surgical and medical procedures) | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 1
Spinal decompression (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 2 | 3
Spinal laminectomy (Surgical and medical procedures) | 1 | 3
Stent placement (Surgical and medical procedures) | 2 | 2
Surgery (Surgical and medical procedures) | 1 | 2
Thalamotomy (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 1 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 2
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 3 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 6
Embolism (Vascular disorders) | 0 | 1
Fibromuscular dysplasia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 2 | 3
Thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=867) | Creatine (N=874)
Cataract (Eye disorders) | 51 | 44
Constipation (Gastrointestinal disorders) | 107 | 121
Diarrhoea (Gastrointestinal disorders) | 50 | 65
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 53 | 39
Nausea (Gastrointestinal disorders) | 101 | 99
Fatigue (General disorders) | 47 | 48
Oedema (General disorders) | 139 | 154
Pain (Gastrointestinal disorders) | 122 | 121
Sinusitis (Infections and infestations) | 46 | 55
Upper respiratory tract infection (Infections and infestations) | 63 | 66
Urinary tract infection (Infections and infestations) | 109 | 85
Fall (Injury, poisoning and procedural complications) | 97 | 91
Weight decreased (Investigations) | 50 | 35
Weight increased (Investigations) | 101 | 137
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 81
Back pain (Musculoskeletal and connective tissue disorders) | 106 | 105
Muscle spasms (Musculoskeletal and connective tissue disorders) | 53 | 101
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 45 | 43
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 47
Dizziness (Nervous system disorders) | 81 | 62
Somnolence (Nervous system disorders) | 67 | 61
Anxiety (Psychiatric disorders) | 77 | 65
Depression (Psychiatric disorders) | 106 | 100
Hallucination (Psychiatric disorders) | 39 | 45
Insomnia (Psychiatric disorders) | 101 | 96
Pollakiuria (Renal and urinary disorders) | 50 | 34
Proteinuria (Renal and urinary disorders) | 49 | 47
Hypertension (Vascular disorders) | 46 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No